CLINICAL TRIAL: NCT04751409
Title: Evaluating the Impact of Limited vs. Intense Post-Operative Surveillance on Patient-Reported Outcomes in Patients With Soft Tissue Sarcoma
Brief Title: Evaluating the Impact of Limited Compared With Intense Post-Operative Surveillance on Patient-Reported Outcomes in Patients With Stage II-III Soft Tissue Sarcoma of the Trunk and Extremities
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0854; NCI-2021-00436 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0854 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Stage II Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage III Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IIIA Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IIIB Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8
MeSH Terms: interventions — X-Rays; Chromatin Immunoprecipitation Sequencing; Follow-Up Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1, Arm I (intense follow up) (Experimental): Patients undergo intense follow-up every 3 months for 2 years consisting of restaging with CT-chest and imaging of the primary site.
  Interventions: Procedure: Computed Tomography; Procedure: Follow-Up; Procedure: Imaging Technique; Other: Questionnaire Administration
- Group 1, Arm II (limited follow-up) (Experimental): Patients undergo limited follow-up every 6 months for 2 years consisting of restaging with either CT-chest or CXR and imaging of the primary site.
  Interventions: Procedure: Chest Radiography; Procedure: Computed Tomography; Procedure: Follow-Up; Procedure: Imaging Technique; Other: Questionnaire Administration
- Group 2 (intense follow up) (Experimental): Patients undergo intense follow-up every 3 months for 2 years as in Group 1, Arm I.
  Interventions: Procedure: Computed Tomography; Procedure: Follow-Up; Procedure: Imaging Technique; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Chest Radiography — Undergo CXR
  Other Names: Chest X-ray
  Arms: Group 1, Arm II (limited follow-up)
Procedure: Computed Tomography — Undergo CT-chest
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Follow-Up — Undergo intense follow-up
  Other Names: Active Follow-up; Clinical Signs Follow-up; CLSFUP; Follow Up; follow_up; Followed; Followup
  Arms: Group 1, Arm I (intense follow up); Group 2 (intense follow up)
Procedure: Follow-Up — Undergo limited follow-up
  Other Names: Active Follow-up; Clinical Signs Follow-up; CLSFUP; Follow Up; follow_up; Followed; Followup
  Arms: Group 1, Arm II (limited follow-up)
Procedure: Imaging Technique — Undergo imaging
  Other Names: Diagnostic Imaging Technique; Imaging; imaging procedure; Imaging Procedures; Imaging, Not Otherwise Specified; Medical Imaging
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how anxiety is affected by 2 types of follow-up after surgery, limited follow-up and intense follow-up, in patients with stage II-III soft tissue sarcoma of the trunk and extremities. In cancer survivors, the fear of cancer coming back (recurring) is common and may persist long after the end of treatment. It may also be exacerbated by return visits for imaging (surveillance). The purpose of this study is to determine how patients' anxiety and other cancer-related outcomes are affected by how often surveillance is done.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether a risk-based limited follow-up surveillance is associated with reduced patient anxiety compared to risk-based intense surveillance.

SECONDARY OBJECTIVE:

I. To evaluate the impact of reduced surveillance in low-risk patients on overall survival, time to local or distant recurrence, anxiety at early and late time-points, out of pocket costs, and number of missed or extra clinic visits, compared to the risk-based intense follow-up in both low-risk and high-risk patients.

OUTLINE: Patients are assigned to 1 of 2 groups based on risk status.

GROUP 1 (LOW RISK): Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo intense follow-up every 3 months for 2 years consisting of restaging with computed tomography (CT)-chest and imaging of the primary site.

ARM II: Patients undergo limited follow-up every 6 months for 2 years consisting of restaging with either CT-chest or chest x-ray (CXR) and imaging of the primary site.

GROUP 2 (HIGH RISK): Patients undergo intense follow-up every 3 months for 2 years as in Group 1, Arm I.

ELIGIBILITY:
IInclusion Criteria:

* ≥18 years old
* Completion of sarcoma therapy (chemotherapy, radiation therapy and/or surgery) within 8-14 weeks of study enrollment
* Willingness to complete surveys x 2 years

Exclusion Criteria:

* Documented metastatic disease at the time of enrollment
* Non-English-speaking patients

Pregnant women will be included in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Estimated)
Dates: Start 2020-12-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Total score for Fear of Cancer Recurrence Inventory - Short Form | Baseline to 12 months after surgery
  Will be calculated as the area under the curve by obtaining patient-reported outcomes at 4 separate time points and then graphically calculating and comparing the area under the curve for each patient. The mean area under the curve of the Fear of Cancer Recurrence Inventory - Short Form will be estimated along with a 95% confidence interval within each study group.
Mean area under the curve of the Fear of Cancer Recurrence Inventory - Short Form | Up to 12 months after surgery
  Will be estimated along with a 95% confidence interval within each study group.

SECONDARY OUTCOMES:
Change in fear of recurrence | Baseline up to 24 months post-resection
  Will be assessed by the Fear of Cancer Recurrence Inventory - Short Form via linear mixed models over time and to compare changes of these assessments over time between the two low-risk groups adjusting for important covariates such age, gender and other patient prognostic factors.
Change in distress | Baseline up to 24 months post-resection
  Will be assessed by the Impact of Events scale via linear mixed models over time and to compare changes of these assessments over time between the two low-risk groups adjusting for important covariates such age, gender and other patient prognostic factors.
Change in anxiety and depression | Baseline up to 24 months post-resection
  Will be assessed by the Hospital Anxiety and Depression Scale via linear mixed models over time and to compare changes of these assessments over time between the two low-risk groups adjusting for important covariates such age, gender and other patient prognostic factors.
Change in out-of-pocket costs | Baseline up to 24 months post-resection
  Will be assessed by the Cost Survey via linear mixed models over time and to compare changes of these assessments over time between the two low-risk groups adjusting for important covariates such age, gender and other patient prognostic factors.
Time to local recurrence | From time of surgery to local recurrence as defined by Response Evaluation Criteria in Solid Tumors (RECIST) or death from any cause, whichever occurs first, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in survival between groups.
Time to distant metastasis | From time of surgery to distant metastasis as defined by RECIST or death from any cause, whichever occurs first, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in survival between groups.
Overall survival | From time of surgery to death, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in survival between groups.
Number of missed or extra clinic visits | Up to 2 years
  The analysis of number of missed or extra clinic visits will be descriptive in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Roland, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org